CLINICAL TRIAL: NCT00000553
Title: HDL-Atherosclerosis Treatment Study (HATS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Factorial | Purpose: Prevention
Other Study IDs: 97; R01HL049546 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Simvastatin; Niacin; Antioxidants

INTERVENTIONS:
Drug: simvastatin
Drug: niacin
Drug: antioxidants

SUMMARY:
To measure the effects of lipid-lowering drugs and/or antioxidant vitamins on progression or regression of coronary heart disease as measured by quantitative angiography in patients with low high density lipoprotein (HDL) cholesterol.

DETAILED DESCRIPTION:
BACKGROUND:

More than one-third of patients with coronary disease have "low" high density lipoprotein cholesterol (HDLc) levels (less than 35 mg/dl; United States 20th percentile) and "normal" low density lipoprotein cholesterol (LDLc) (less than 145; United States mean), a group for whom current treatment guidelines are not based on clinical trial data. Low HDLc levels are strong, independent predictors of cardiovascular disease and cardiovascular mortality risk, equally so for both men and women. This high coronary artery disease risk may be due to an imbalance between delivery of cholesterol into the arterial intima by LDL and its removal by HDL. Also, since HDL serve as antioxidants and cytoprotectants, an important HDL role may be to prevent LDL oxidation and thus limit macrophage-mediated intimal lipid accumulation or to prevent vascular cell toxicity. Recent epidemiologic, experimental, and clinical trial evidence suggests that a 15 mg/dl rise in HDL cholesterol would reduce coronary artery disease incidence and mortality by 30 to 70 percent and that antioxidant vitamins E, C, and beta-carotene might reduce coronary artery disease events and atherogenesis. The potential absolute benefit is much greater in those with existing coronary artery disease. It has also been shown that HDLc rises in response to exercise, smoking cessation, weight reduction, and monounsaturated fats.

DESIGN NARRATIVE:

Randomized, Phase III. Each patient was randomly assigned to a lipid-altering strategy or its placebo and to an antioxidant vitamin strategy or its placebo, in a 2 x 2 factorial design. The four groups were simvastatin-niacin plus an antioxidant vitamin cocktail; simvastatin-niacin plus vitamin placebo; antioxidant vitamins alone plus simvastatin-niacin placebo; or placebos for both strategies. All groups were counseled with respect to diet, exercise, and smoking cessation. The primary endpoint was the average change in proximal obstructive disease during the 2.5 year interval between baseline and the followup study. Secondary endpoints included the frequency of cardiac events, including cardiac death, confirmed non-fatal myocardial infarction, cerebrovascular accident, or revascularization by bypass or angioplasty for medically refractory unstable ischemia. The trial ended in August, 1999.

ELIGIBILITY:
Men and women with low HDL cholesterol, with at least one 50% stenotic coronary lesion or three 30% stenotic coronary lesions. Women range in age from 35 to less than 68 and men from 35 to less than 63.

Ages: 35 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1994-09; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Brown — University of Washington

REFERENCES:
- [Background] Brown G, Stewart BF, Zhao XQ, Hillger LA, Poulin D, Albers JJ. What benefit can be derived from treating normocholesterolemic patients with coronary artery disease? Am J Cardiol. 1995 Sep 28;76(9):93C-97C. doi: 10.1016/s0002-9149(99)80477-9. PMID 7572694
- [Background] Brown BG, Zhao XQ, Chait A, Frohlich J, Cheung M, Heise N, Dowdy A, DeAngelis D, Fisher LD, Albers J. Lipid altering or antioxidant vitamins for patients with coronary disease and very low HDL cholesterol? The HDL-Atherosclerosis Treatment Study Design. Can J Cardiol. 1998 Apr;14 Suppl A:6A-13A. PMID 9594927
- [Background] Cheung MC, Wolfbauer G, Brown BG, Albers JJ. Relationship between plasma phospholipid transfer protein activity and HDL subclasses among patients with low HDL and cardiovascular disease. Atherosclerosis. 1999 Jan;142(1):201-5. doi: 10.1016/s0021-9150(98)00190-7. PMID 9920522
- [Background] Brown BG, Zhao XQ, Chait A, Fisher LD, Cheung MC, Morse JS, Dowdy AA, Marino EK, Bolson EL, Alaupovic P, Frohlich J, Albers JJ. Simvastatin and niacin, antioxidant vitamins, or the combination for the prevention of coronary disease. N Engl J Med. 2001 Nov 29;345(22):1583-92. doi: 10.1056/NEJMoa011090. PMID 11757504
- [Background] Brown BG, Cheung MC, Lee AC, Zhao XQ, Chait A. Antioxidant vitamins and lipid therapy: end of a long romance? Arterioscler Thromb Vasc Biol. 2002 Oct 1;22(10):1535-46. doi: 10.1161/01.atv.0000034706.24149.95. PMID 12377728
- [Derived] Williams PT, Zhao XQ, Marcovina SM, Otvos JD, Brown BG, Krauss RM. Comparison of four methods of analysis of lipoprotein particle subfractions for their association with angiographic progression of coronary artery disease. Atherosclerosis. 2014 Apr;233(2):713-720. doi: 10.1016/j.atherosclerosis.2014.01.034. Epub 2014 Jan 30. PMID 24603218
- [Derived] Williams PT, Zhao XQ, Marcovina SM, Brown BG, Krauss RM. Levels of cholesterol in small LDL particles predict atherosclerosis progression and incident CHD in the HDL-Atherosclerosis Treatment Study (HATS). PLoS One. 2013;8(2):e56782. doi: 10.1371/journal.pone.0056782. Epub 2013 Feb 27. PMID 23460815